CLINICAL TRIAL: NCT01638949
Title: Study of the Predictive Markers and the Pathophysiological Mechanisms of Alzheimer's Disease: Transverse and Longitudinal Approach in Anatomical and Functional Multimodal Imaging
Brief Title: Multi-modal Neuroimaging in Alzheimer's Disease
Acronym: IMAP+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-A01493-38
Record Dates: First submitted 2012-05-22; First posted 2012-07-12 (Estimated); Last update posted 2023-12-07 (Actual); Status verified 2014-04

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; MCI; genetic; AV45-PET
MeSH Terms: conditions — Alzheimer Disease | interventions — Apolipoprotein E4

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Young controls (Experimental)
  Interventions: Behavioral: Memory assessment; Biological: Circulating biomarkers measure; Genetic: ApoE4; Other: Brain imaging examination MRI and PET examinations
- Middle age controls (Experimental)
  Interventions: Behavioral: Memory assessment; Biological: Circulating biomarkers measure; Genetic: ApoE4; Other: Brain imaging examination MRI and PET examinations
- Elderly controls (Experimental)
  Interventions: Behavioral: Memory assessment; Biological: Circulating biomarkers measure; Genetic: ApoE4; Other: Brain imaging examination MRI and PET examinations
- Asymptomatic subjects (Experimental): Asymptomatic subjects from families carrying a genetic mutation with an autosomal dominant transmission
  Interventions: Behavioral: Memory assessment; Biological: Circulating biomarkers measure; Genetic: ApoE4; Other: Brain imaging examination MRI and PET examinations
- Subjectif Cognitive Impariment patients (Experimental)
  Interventions: Behavioral: Memory assessment; Biological: Circulating biomarkers measure; Genetic: ApoE4; Other: Brain imaging examination MRI and PET examinations
- Mild Cognitive Impairment patients (Experimental)
  Interventions: Behavioral: Memory assessment; Biological: Circulating biomarkers measure; Genetic: ApoE4; Other: Brain imaging examination MRI and PET examinations
- Alzheimer Disease patients (Experimental)
  Interventions: Behavioral: Memory assessment; Biological: Circulating biomarkers measure; Genetic: ApoE4; Other: Brain imaging examination MRI and PET examinations
- Non degenerative amnsesic syndrome (Experimental)
  Interventions: Behavioral: Memory assessment; Biological: Circulating biomarkers measure; Genetic: ApoE4; Other: Brain imaging examination MRI and PET examinations

INTERVENTIONS:
Behavioral: Memory assessment — Neuropsycological tests including clinical and original tests to compare differences between each populations.
Biological: Circulating biomarkers measure — ELISA tests from blood samples to compare differences between each populations.
Genetic: ApoE4 — Evaluation of apolipoprotein E polymorphism as a risk factor.
Other: Brain imaging examination MRI and PET examinations — Structural and functional MRI FDG-PET to compare differences between each populations.

SUMMARY:
Alzheimer's disease (AD) is a major public health problem due to its socio-economic weight. An early diagnosis of AD is urgently needed as it would constitute a determinant breakthrough from a social, financial and research standpoints. Therefore, the investigators need predictive markers of AD, and neuroimaging is a particularly promising tool, especially when using complementary neuroimaging techniques and a longitudinal design, allowing to assess the relationships between the different biomarkers of the disease, their dynamic and their chronology.

DETAILED DESCRIPTION:
The three main objectives of this project are:

* To Identify, compare and combine the predictive markers of AD,
* To better understand the pathophysiologic mechanisms of AD,
* To study the ability of different neuroimaging techniques to monitor AD's evolution.

For these purposes, detailed neuropsychological evaluations, biological measures and brain structural & functional imaging measures are associated for a fully-comprehensive description of the different manifestations of AD through disease progression and toward identifying early markers.

Subjects are evaluated using neuropsychological tests of episodic memory (encoding vs. retrieval), executive functions (inhibition, flexibility, and updating processes), self-judgment, theory of mind, mental imagery and verbal fluency. A FDG-PET measure of resting state glucose consumption, an AV45-PET measure of amyloid deposition as well as anatomical, resting-state and activation fMRI scans are performed for each volonteer. In addition, blood and cerebro-spinal fluid samples will be performed to determine different biomarkers (Aβ1-40, Aβ1-42 and tPA as circulating blood proteins and Aβ40, Aβ42, tau and its phosphorylated form in CSF). The investigators also study the polymorphism of Apolipoprotein E as a genetic risk factor of AD.

One hundred and twenty healthy controls (40 young, 40 middle age and 40 elderly), 40 Mild Cognitive Impairment patients (MCI; i.e. isolated memory impairment and increased risk of developing AD) and 30 AD patients will be selected. Participants with increased risk of developing AD and without objective evidence will be also studied: 50 asymptomatic subjects from families carrying a genetic mutation with an autosomal dominant transmission (NORMA) and 40 Subjective Cognitive Impairment patients (SCI).

Clinical follow-up of patients will be completed during 36 months (18 months for AD patients), as a neuropsychological evaluation every 6 months. Comparable neuropsychological and imaging exams will be proposed once again after 18 months for all participants as well as after 36 months for elderly controls, NORMA and SCI & MCI patients.

To study and compare the effectiveness of different in vivo markers (to predict cognitive decline in populations at risk of developing AD), each data set (i.e. modality) will be first analyzed independently from one another (intra-modality analyses), including inter-group comparisons, correlations and connectivity analyses, as well as longitudinal assessment of cognitive, biological and brain changes. Baseline data will also be analyzed in function of patient's clinical evolution to assess their predictive value. Comparisons and correlations between the different patterns of alterations will then be performed through inter-modality analyses. More specifically, the investigators will address the questions of the relationships between cognitive and cerebral alterations and structural / functional brain changes over our different patient samples, neuroimaging data sets, and through disease evolution.

This project is expected to identify specific and early markers of the MA and also to compare the diagnostic efficiency of different measures. It should contribute to better understand brain and cognitive alterations in AD. Finally, the investigators will be able to appreciate the dynamic properties of these alterations in the evolution of the disease through the longitudinal study.

ELIGIBILITY:
Inclusion Criteria :

* Education level > 7 years
* Native language: French
* Medical, neurological, neuropsychological and neuroradiological depth in accordance with the criteria for inclusion and exclusion-specific population, that is to say:

  * Healthy young volunteers: between 18 and 40 years old; normal performances compared to the age and the educational level for all tests of the diagnostic battery (± 1.65 SD).
  * Healthy Middle-aged volunteers: between 40 and 60 years old; without memory complaints, normal performances compared to the age and the educational level for all tests of the diagnostic battery (± 1.65 SD).
  * Healthy Elderly volunteers: over 60 years old, living at home, without memory complaints, normal performances compared to the age and the educational level for all tests of the diagnostic battery (± 1.65 SD).
  * SCI patients: over 60 years old ; memory complaints; memory complaint ; normal performances compared to the age and the educational level for all tests of the diagnostic battery (± 1.65 SD).
  * MCI patients: presenting the current criteria for amnestic MCI including: i) memory complaint, ii) deficits of the episodic memory (lower performance of at least 1.65 SD from the norm for age and cultural level for one or more scores of episodic memory and iii) normal performances compared to the age and the educational level of all other cognitive functions as memory, including tests to assess cognitive abilities.
  * Alzheimer's patients: presenting the standard criteria of NINCDS-ADRDA probable Alzheimer's disease, including abnormal global cognitive function and deficits in at least two cognitive domains identified by the diagnostic battery and a mild to moderate Alzheimer's disease (MMSE ≥ 15).

Exclusion Criteria :

* The sudden onset of cognitive impairments (as opposed to their slow and gradual installation in Alzheimer's disease)
* A chronic neurological, psychiatric, endocrine, hepatic or infectious complaint
* A history of major disease (an uncontrolled diabetes, a lung, heart, metabolic, hematologic, endocrine disease or a severe cancer)
* A medication that may interfere with memory or metabolic measures
* A alcohol or drugs abuse
* The cons-indications to MRI (claustrophobia, metallic object in the body)
* A predominantly left-hand (score below 50% in Edinburgh Inventory)
* Protected adults, and persons not affiliated with a social security system will not participate in this study
* The inclusion of a participant in another biomedical research protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Rate of volume change of whole brain, hippocampus and other structural MRI measures | 3 years
Rate of Decline as measured by: Cognitive Tests, Activities of Daily Living, and CDR Sum of Boxes | 3 years
Rates of change on each specified biochemical biomarker | 3 years
Rates of change of glucose metabolism (FDG-PET) | 3 years
Extent of amyloid deposition as measured by 18F-AV45 | 3 years
Group differences for each imaging and biomarker measurement | 3 years
APOE genotype | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Vincent de La Sayette, MD, Principal Investigator — University Hospital, Caen
Locations (7):
- France (7):
  - GIP Cyceron, Caen, Calvados
  - Inserm - EPHE - University of Caen U1077, Caen
  - University Hospital Côte de Nacre, Caen
  - University Hospital Roger Salengro, Lille
  - University Hospital Pontchaillou, Rennes
  - University Hospital Rouen, Rouen
  - University Hospital Tours, Tours

REFERENCES:
- [Derived] Kuhn E, Perrotin A, La Joie R, Touron E, Dautricourt S, Vanhoutte M, Vivien D, de La Sayette V, Chetelat G; Alzheimer's Disease Neuroimaging Initiative. Association of the Informant-Reported Memory Decline With Cognitive and Brain Deterioration Through the Alzheimer Clinical Continuum. Neurology. 2023 Jun 13;100(24):e2454-e2465. doi: 10.1212/WNL.0000000000207338. Epub 2023 Apr 21. PMID 37085328
- [Derived] Kuhn E, Moulinet I, Perrotin A, La Joie R, Landeau B, Tomadesso C, Bejanin A, Sherif S, De La Sayette V, Desgranges B, Vivien D, Poisnel G, Chetelat G. Cross-sectional and longitudinal characterization of SCD patients recruited from the community versus from a memory clinic: subjective cognitive decline, psychoaffective factors, cognitive performances, and atrophy progression over time. Alzheimers Res Ther. 2019 Jul 8;11(1):61. doi: 10.1186/s13195-019-0514-z. PMID 31286994
- [Derived] Gonneaud J, Arenaza-Urquijo EM, Fouquet M, Perrotin A, Fradin S, de La Sayette V, Eustache F, Chetelat G. Relative effect of APOE epsilon4 on neuroimaging biomarker changes across the lifespan. Neurology. 2016 Oct 18;87(16):1696-1703. doi: 10.1212/WNL.0000000000003234. Epub 2016 Sep 28. PMID 27683850